CLINICAL TRIAL: NCT01307436
Title: A Phase III Randomised, Open, Controlled Study to Assess the Safety and Immunogenicity of Concomitant Administration of Virosomal Hepatitis A Vaccine (Epaxal®) With DTPaHibIPV, OPV and MMR Vaccines vs. Non-concomitant Administration in 12-15 Month Old Children. Follow-up: Serological Long-term Follow-up of Subjects for up to 42 Months, 5.5 and 7.5 Years After the Second Dose.
Brief Title: Long Term Follow-up of a Study to Assess the Safety and Immunogenicity of a Hepatitis A Vaccine Administered With and in the Absence of DTPaHibIPV, OPV and MMR Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR106637; EPA 004 FU (Other: Crucell Holland BV)
Record Dates: First submitted 2011-02-28; First posted 2011-03-03 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis A
Keywords: Hepatitis A Vaccine; Combined Vaccines; DTP Vaccine; MMR Vaccine
MeSH Terms: conditions — Hepatitis A; Hepatitis | interventions — epaxal berna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Epaxal + concomitant administration of DTPaHibIPV, MMR, OPV
  Interventions: Biological: Epaxal
- Group B (Experimental): Epaxal, with administration of DTPaHibIPV, MMR, OPV one month later
  Interventions: Biological: Epaxal
- Group C (Active Comparator): Havrix 720 + concomitant administration of DTPaHibIPV, MMR
  Interventions: Biological: Havrix 720

INTERVENTIONS:
Biological: Epaxal — 0.25ml Epaxal: at least 12 IU hepatitis A antigen coupled to immunopotentiating reconstituted influenza virosomes (IRIV)
  Arms: Group A; Group B
Biological: Havrix 720 — 0.5ml Havrix 720: at least 720 EU hepatitis A antigen adsorbed onto aluminium hydroxide
  Arms: Group C

SUMMARY:
The primary purpose of this study was to assess whether the protection afforded by Epaxal vaccine co-administered with diphtheria, tetanus, Bordetella pertussis, Haemophilus influenzae type b, and inactivated polio vaccine(DTPaHibIPV), oral polio vaccine (OPV) and (measles mumps and rubella) MMR vaccines against hepatitis A was not inferior to the protection afforded by Epaxal administered alone. The aim of the follow-up phase is to obtain information on the long term protection afforded by Epaxal, and to compare this with an alternative hepatitis A vaccine (Havrix).

ELIGIBILITY:
Inclusion Criteria:

Original study:

* Written informed consent obtained from the parent/legal guardian of the subject.
* Free of obvious health problems as established by medical history and/or clinical examination before entering the study.
* At least 8 kg of body weight at age of 12 months.

Follow-up phase:

* Subjects enrolled and randomised in the original study and having received two doses of the hepatitis A study vaccines.

Exclusion Criteria:

Original study:

* Children not having received 3 documented doses of DTPaHib and polio vaccines during infancy
* Children having received a documented dose of MMR during infancy
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and the 30 days safety follow-up after the last dose.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of systemic corticosteroids (inhaled and topical steroids are allowed).
* Administration of a vaccine not foreseen by the study protocol within 4 weeks prior to the first dose of study vaccine.
* Previous vaccination against hepatitis A.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness
* Acute disease at the time of enrolment.

Follow-up phase:

* Children who had received a hepatitis A antigen containing vaccine since the last visit

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 327 (Actual)
Dates: Start 2007-03-14 (Actual); Primary Completion 2013-07-08 (Actual); Study Completion 2013-07-08 (Actual)

PRIMARY OUTCOMES:
Anti-hepatitis A virus (HAV) antibody concentrations | 5.5 years
  Individual anti-HAV antibody concentrations determined by enzyme-linked immunosorbent assay
Anti-hepatitis A virus (HAV) antibody concentrations | 7.5 years
  Individual anti-HAV antibody concentrations determined by enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Geometric mean concentrations (GMC) | 5.5 and 7.5 years
  GMCs of anti-HAV antibodies
Proportion of seroprotected subjects | 5.5 and 7.5 years
  Proportion of subjects seroprotected defined as anti-HAV antibody concentrations of at least 10 mIU/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ron Dagan, MD, Principal Investigator — Soraka Medical Center; Shai Ashkenazi, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (2):
- Israel (2):
  - Beersheba
  - Petah Tikva

REFERENCES:
- [Result] Dagan R, Ashkenazi S, Livni G, Go O, Bagchi P, Sarnecki M. Long-term Serologic Follow-up of Children Vaccinated with a Pediatric Formulation of Virosomal Hepatitis A Vaccine Administered With Routine Childhood Vaccines at 12-15 Months of Age. Pediatr Infect Dis J. 2016 Jul;35(7):e220-8. doi: 10.1097/INF.0000000000001176. PMID 27093164